CLINICAL TRIAL: NCT04283942
Title: Effect of Intermittent Calorie Restriction on Metabolic Dysfunction-Associated Steatotic Liver Disease Patients With Abnormal Glucose Metabolism
Brief Title: Effect of Intermittent Calorie Restriction on MASLD Patients With Abnormal Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hua Bian, Director, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-256R
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Fatty Liver Disease; Type 2 Diabetes; Impaired Glucose Regulation
Keywords: Metabolic dysfunction-associated steatotic liver disease; Type 2 Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into intermittent calorie restriction group and control group for 12 weeks of intervention. Both groups will be followed up 4 weeks after intervention.
  ICR group: during the 2-day fasting-mimicking period each week, the food based on plant ingredients will be served (4 pieces of nutrition bars / day, 1:2:1 for breakfast, lunch and dinner, 124.4kcal/piece, 497.2kcal / day in total). In the rest 5 days each week, subjects are allowed ad libitum to their usual food.
  Control group: continuous calorie restriction (CCR). Under the guidance of nutritionist, subjects have to learn the method of food calories calculation. For each day, the daily calories intake is limited to 25 kcal / kg × standard weight [kg, estimated by height (cm) - 100].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Calorie Restriction (ICR) (Experimental): Participants in ICR group were instructed to ensure 2 successive days of fasting-mimicking and 5 days of recovery per week. On fasting-mimicking days, the participants were instructed to consume approximately 500 kcal/day and they were provided with plant-based meal replacement (ZhenBaiNian nutrition bar, Beijing Wanlaikang Nutrition and Health Food Science and Technology Research Institute Co., Ltd, China) to improve adherence and ensured adequate intake of micronutrients. In the rest 5 days of recovery per week, participants were allowed to consume their usual diet.
  Interventions: Behavioral: Intermittent calorie restriction (ICR)
- Control (Continuous calorie restriction, CCR) (Other): Participants in control group were instructed to consume the prescribed calories (25 kcal / kg × [height (cm) - 100] kg) every day by eating conventional food without time restriction.
  Interventions: Behavioral: Continuous calorie restriction (CCR)

INTERVENTIONS:
Behavioral: Intermittent calorie restriction (ICR) — Participants in ICR group were instructed to ensure 2 successive days of fasting-mimicking and 5 days of recovery per week. On fasting-mimicking days, the participants were instructed to consume approximately 500 kcal/day and they were provided with plant-based meal replacement to improve adherence and ensured adequate intake of micronutrients. In the rest 5 days of recovery per week, participants were allowed to consume their usual diet.
  Participants will receive dietary counseling from experienced nutritionists and eat a balanced diet (macronutrient distribution of approximately 10-15% protein, 55-65% carbohydrate and 20-30% fat).They are required to write daily dietary log. Besides, they are required to maintain their exercise routines and record their daily steps using a unified pedometer (Redmi Smart Band, Xiaomi Corporation, China). The use of drugs affecting blood glucose and LFC will be avoided.
  Other Names: Intermittent fasting
  Arms: Intermittent Calorie Restriction (ICR)
Behavioral: Continuous calorie restriction (CCR) — Participants in CCR group were instructed to consume the prescribed calories (25 kcal / kg × [height (cm) - 100] kg) every day by eating conventional food without time restriction.
  Participants will receive dietary counseling from experienced nutritionists and eat a balanced diet (macronutrient distribution of approximately 10-15% protein, 55-65% carbohydrate and 20-30% fat).They are required to write daily dietary log. Besides, they are required to maintain their exercise routines and record their daily steps using a unified pedometer (Redmi Smart Band, Xiaomi Corporation, China). The use of drugs affecting blood glucose and LFC will be avoided.
  Other Names: Daily calorie restriction
  Arms: Control (Continuous calorie restriction, CCR)

SUMMARY:
This study is designed to observe the effect of 5:2 intermittent calorie restriction (fasting 2 days each week) on liver fat content in MASLD patients with abnormal blood glucose.

DETAILED DESCRIPTION:
Intermittent caloric restriction (ICR) can effectively reduce weight and facilitate blood glucose control, but whether it can be applied for clinical treatment to metabolic dysfunction-associated steatotic liver disease (MASLD) patients remains unclear. We intend to carry out this study in MASLD patients with abnormal glucose metabolism. It is an open-labeled randomized trial designed to observe the effect of 5:2 intermittent calorie restriction (fasting 2 days each week) on liver fat content in MASLD patients with abnormal blood glucose. 60 patients will be randomly divided into ICR group and control group for 12 weeks of intervention. ICR group: during the 2-day fasting-mimicking period each week, the food based on plant ingredients will be served (4 pieces of nutrition bars / day, 1:2:1 for breakfast, lunch and dinner, 124.4kcal / piece, 497.2kcal / day in total). In the rest 5 days each week, subjects are allowed ad libitum to their usual food. Control group (continuous calorie restriction, CCR): under the guidance of nutritionist, subjects have to learn the method of food calories calculation. The daily calories intake for control group should be: 25 kcal / kg × [height (cm) - 100] kg. Daily food diary is required in both groups. During the experiment, all subjects should maintain their exercise routine. The use of drugs affecting blood glucose and fatty liver should be avoided. After 12 weeks of intervention, the changes of liver fat content were evaluated by magnetic resonance spectroscopy (MRS) and Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF). The effects of ICR on body weight, blood glucose and body fat will also be evaluated. Both groups will be followed up on their changes of weight 4 weeks after intervention.

ELIGIBILITY:
Inclusion Criteria

* Age 18-70
* Diagnosed as fatty liver by ultrasound or magnetic resonance imaging
* BMI ≥ 24 kg/m2
* abnormal glucose metabolism: (meeting at least one):

  1. Impaired glucose regulation: fasting blood glucose ≥ 100 mg/dL, postprandial blood glucose ≥ 140 mg/dL or HbA1c ≥ 5.7%
  2. Diabetes mellitus: diabetic symptoms + plasma glucose concentration ≥ 200 mg/dL at any time or fasting plasma glucose concentration ≥ 100 mg/dL or OGTT 2 h plasma glucose concentration ≥ 200 mg/dL

Exclusion Criteria

* Type 1 diabetes, gestational diabetes and other special types of diabetes
* Poor blood glucose control, HbA1c > 8.5% within 3 months
* Taking antidiabetic drugs in the past month
* Serum ALT > 6 times of normal upper limit
* Excessive alcohol consumption (alcohol intake: men > 140 g, women > 70 g in the past 6 months)
* Other liver diseases: such as acute and chronic viral hepatitis, drug-induced hepatitis, immune hepatitis, liver cirrhosis, liver cancer, etc
* Taking drugs that may affect MASLD in the past three months, such as vitamin E
* Biliary obstructive diseases
* Other diseases affecting glucose and lipid metabolism: hyperthyroidism, hypothyroidism, Cushing's syndrome, etc
* Chronic kidney disease (serum creatinine ≥ 2.0 mg/dL)
* Life expectancy of no more than 5 years
* Already pregnant or plan to be pregnant in the near future
* Mental illness
* Other conditions affecting follow-up
* Have participated in other clinical trials in the past 4 weeks
* Absent of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hua Bian, Principal Investigator — Shanghai Zhongshan Hospital; Xin Gao, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Fan JG, Kim SU, Wong VW. New trends on obesity and NAFLD in Asia. J Hepatol. 2017 Oct;67(4):862-873. doi: 10.1016/j.jhep.2017.06.003. Epub 2017 Jun 19. PMID 28642059
- [Background] Fan JG. Epidemiology of alcoholic and nonalcoholic fatty liver disease in China. J Gastroenterol Hepatol. 2013 Aug;28 Suppl 1:11-7. doi: 10.1111/jgh.12036. PMID 23855290
- [Background] Wang FS, Fan JG, Zhang Z, Gao B, Wang HY. The global burden of liver disease: the major impact of China. Hepatology. 2014 Dec;60(6):2099-108. doi: 10.1002/hep.27406. Epub 2014 Oct 29. PMID 25164003
- [Background] Angulo P. Nonalcoholic fatty liver disease. N Engl J Med. 2002 Apr 18;346(16):1221-31. doi: 10.1056/NEJMra011775. No abstract available. PMID 11961152
- [Background] Ballestri S, Zona S, Targher G, Romagnoli D, Baldelli E, Nascimbeni F, Roverato A, Guaraldi G, Lonardo A. Nonalcoholic fatty liver disease is associated with an almost twofold increased risk of incident type 2 diabetes and metabolic syndrome. Evidence from a systematic review and meta-analysis. J Gastroenterol Hepatol. 2016 May;31(5):936-44. doi: 10.1111/jgh.13264. PMID 26667191
- [Background] Vozarova B, Stefan N, Lindsay RS, Saremi A, Pratley RE, Bogardus C, Tataranni PA. High alanine aminotransferase is associated with decreased hepatic insulin sensitivity and predicts the development of type 2 diabetes. Diabetes. 2002 Jun;51(6):1889-95. doi: 10.2337/diabetes.51.6.1889. PMID 12031978
- [Background] Armstrong MJ, Adams LA, Canbay A, Syn WK. Extrahepatic complications of nonalcoholic fatty liver disease. Hepatology. 2014 Mar;59(3):1174-97. doi: 10.1002/hep.26717. Epub 2014 Jan 16. PMID 24002776
- [Background] Musso G, Gambino R, Tabibian JH, Ekstedt M, Kechagias S, Hamaguchi M, Hultcrantz R, Hagstrom H, Yoon SK, Charatcharoenwitthaya P, George J, Barrera F, Hafliethadottir S, Bjornsson ES, Armstrong MJ, Hopkins LJ, Gao X, Francque S, Verrijken A, Yilmaz Y, Lindor KD, Charlton M, Haring R, Lerch MM, Rettig R, Volzke H, Ryu S, Li G, Wong LL, Machado M, Cortez-Pinto H, Yasui K, Cassader M. Association of non-alcoholic fatty liver disease with chronic kidney disease: a systematic review and meta-analysis. PLoS Med. 2014 Jul 22;11(7):e1001680. doi: 10.1371/journal.pmed.1001680. eCollection 2014 Jul. PMID 25050550
- [Background] Huang MA, Greenson JK, Chao C, Anderson L, Peterman D, Jacobson J, Emick D, Lok AS, Conjeevaram HS. One-year intense nutritional counseling results in histological improvement in patients with non-alcoholic steatohepatitis: a pilot study. Am J Gastroenterol. 2005 May;100(5):1072-81. doi: 10.1111/j.1572-0241.2005.41334.x. PMID 15842581
- [Background] Sundfor TM, Svendsen M, Tonstad S. Intermittent calorie restriction-a more effective approach to weight loss? Am J Clin Nutr. 2018 Nov 1;108(5):909-910. doi: 10.1093/ajcn/nqy288. No abstract available. PMID 30475966
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Background] Cheng CW, Villani V, Buono R, Wei M, Kumar S, Yilmaz OH, Cohen P, Sneddon JB, Perin L, Longo VD. Fasting-Mimicking Diet Promotes Ngn3-Driven beta-Cell Regeneration to Reverse Diabetes. Cell. 2017 Feb 23;168(5):775-788.e12. doi: 10.1016/j.cell.2017.01.040. PMID 28235195
- [Background] Johari MI, Yusoff K, Haron J, Nadarajan C, Ibrahim KN, Wong MS, Hafidz MIA, Chua BE, Hamid N, Arifin WN, Ma ZF, Lee YY. A Randomised Controlled Trial on the Effectiveness and Adherence of Modified Alternate-day Calorie Restriction in Improving Activity of Non-Alcoholic Fatty Liver Disease. Sci Rep. 2019 Aug 2;9(1):11232. doi: 10.1038/s41598-019-47763-8. PMID 31375753
- [Background] Schubel R, Nattenmuller J, Sookthai D, Nonnenmacher T, Graf ME, Riedl L, Schlett CL, von Stackelberg O, Johnson T, Nabers D, Kirsten R, Kratz M, Kauczor HU, Ulrich CM, Kaaks R, Kuhn T. Effects of intermittent and continuous calorie restriction on body weight and metabolism over 50 wk: a randomized controlled trial. Am J Clin Nutr. 2018 Nov 1;108(5):933-945. doi: 10.1093/ajcn/nqy196. PMID 30475957
- [Background] Liu M, Yan HM, Gao X, Gao J. [Association of abnormality of liver enzymes and metabolic syndrome in patients with nonalcoholic fatty liver disease]. Zhonghua Yi Xue Za Zhi. 2007 Jan 23;87(4):253-5. Chinese. PMID 17425870
- [Derived] Sun X, Li F, Yan H, Chang X, Yao X, Yang X, Wu S, Suo Y, Zhu X, Wang C, Gao J, Wang H, Chen Y, Xia M, Bian H, Gao X. Intermittent compared with continuous calorie restriction for treatment of metabolic dysfunction-associated steatotic liver disease: a randomized clinical trial. Am J Clin Nutr. 2025 Jan;121(1):158-166. doi: 10.1016/j.ajcnut.2024.10.012. Epub 2024 Oct 22. PMID 39447676

RESULTS

PARTICIPANT FLOW:
Groups:
- Intermittent Calorie Restriction (ICR): Intermittent calorie restriction (ICR): Participants in ICR group were instructed to ensure 2 successive days of fasting-mimicking and 5 days of recovery per week. On fasting-mimicking days, the participants were instructed to consume approximately 500 kcal/day and they were provided with plant-based meal replacement to improve adherence and ensured adequate intake of micronutrients. In the rest 5 days of recovery per week, participants were allowed to consume their usual diet.
  Participants will receive dietary counseling from experienced nutritionists and eat a balanced diet (macronutrient distribution of approximately 10-15% protein, 55-65% carbohydrate and 20-30% fat). They are required to write daily dietary log. Besides, they are required to maintain their exercise routines and record their daily steps using a unified pedometer (Redmi Smart Band, Xiaomi Corporation, China). The use of drugs affecting blood glucose and LFC will be avoided.
- Control (Continuous Calorie Restriction, CCR): Continuous calorie restriction (CCR): Participants in CCR group were instructed to consume the prescribed calories (25 kcal / kg × [height (cm) - 100] kg) every day by eating conventional food without time restriction.
  Participants will receive dietary counseling from experienced nutritionists and eat a balanced diet (macronutrient distribution of approximately 10-15% protein, 55-65% carbohydrate and 20-30% fat). They are required to write daily dietary log. Besides, they are required to maintain their exercise routines and record their daily steps using a unified pedometer (Redmi Smart Band, Xiaomi Corporation, China). The use of drugs affecting blood glucose and LFC will be avoided.
Period: Overall Study
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (10.7) | 46.5 (11.1) | 47.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 16 | 20 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60
Duration of MASLD [Mean (Standard Deviation); unit: years] | 9.7 (8.8) | 8.6 (7.5) | 9.2 (8.1)
Height [Mean (Standard Deviation); unit: cm] | 165.4 (8.3) | 168.9 (8.8) | 167.2 (8.7)
Weight [Mean (Standard Deviation); unit: kg] | 79.4 (11.4) | 88.6 (19.5) | 84.0 (16.5)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 29.0 (3.2) | 31.1 (5.3) | 30.0 (4.5)
Waist circumference [Mean (Standard Deviation); unit: cm] | 97.6 (7.5) | 100.3 (13) | 98.9 (10.6)
Visceral adipose area [Mean (Standard Deviation); unit: cm2] | 194.4 (56.4) | 195.7 (56.2) | 195.0 (55.8)
Subcutaneous adipose area [Mean (Standard Deviation); unit: cm2] | 315.5 (82.4) | 335.5 (125.2) | 325.4 (105.2)
Lean mass [Mean (Standard Deviation); unit: kg] | 51.5 (10.0) | 57 (12.8) | 54.1 (11.7)
Fat mass [Mean (Standard Deviation); unit: kg] | 27.9 (7.2) | 31.8 (10.1) | 29.8 (8.9)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 135.4 (17.2) | 134.3 (16.6) | 134.8 (16.8)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 82.1 (11.1) | 81.4 (10.2) | 81.8 (10.6)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 115.6 (22.0) | 111.8 (17.1) | 113.8 (19.6)
2h postprandial plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 205.9 (74.2) | 171.2 (79.6) | 188.5 (78.1)
HbA1c [Mean (Standard Deviation); unit: %] | 6.2 (0.8) | 5.9 (0.6) | 6.1 (0.7)
Fasting insulin [Mean (Standard Deviation); unit: μU/mL] | 19.0 (11.8) | 23.5 (15.4) | 21.3 (13.8)
Homeostasis model assessment of insulin resistance (HOMA-IR) index [Mean (Standard Deviation); unit: index] — HOMA-IR index was calculated as fasting serum insulin (μU/ml) × fasting plasma glucose (mmol/l)/22.5. A HOMA-IR index higher than 75th quartile of non diabetes subjects is considered to be insulin resistance. However, due to differences in race, gender and research subjects, there is currently no recognized cut-off point. A study on Caucasian non diabetes population showed that the cut-off value is 2.29. And a Chinese study proposed that the cut-off value of population over 40 years old in Shanghai was 4.31 for men and 4.51 for women.
  index | 5.5 (4.0) | 6.4 (4.2) | 6.0 (4.1)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 182.6 (33.2) | 189.6 (29.7) | 186.1 (31.7)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 152.2 (68.1) | 184.1 (146) | 168.2 (114.2)
HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 44.8 (6.9) | 45.9 (13.9) | 45.3 (10.8)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 107.3 (30.1) | 110.0 (26.6) | 108.9 (28.2)
Free fatty acids [Mean (Standard Deviation); unit: mg/dL] | 17.2 (5.9) | 14.1 (4.8) | 15.5 (5.7)
Alanine aminotransferase [Mean (Standard Deviation); unit: U/L] | 51.5 (38.6) | 37.1 (22.4) | 44.3 (32.1)
Aspartate aminotransferase [Mean (Standard Deviation); unit: U/L] | 32.3 (18.3) | 24.3 (10.2) | 28.3 (15.2)
γ-Glutamyl transpeptidase [Mean (Standard Deviation); unit: U/L] | 39.6 (24.6) | 36.2 (20.3) | 37.9 (22.4)
Liver fat content by 1H-MRS [Mean (Standard Deviation); unit: %] | 37.7 (16.2) | 38.5 (16.1) | 38.1 (16.0)
Liver fat content by Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) [Mean (Standard Deviation); unit: %] — MRI-PDFF is a viable method for the quantification of whole liver and segmental liver fat content. The Couinaud classification is the most widely used system to describe functional liver anatomy.
  1. Caudate
  2. Superior subsegment of the lateral segment
  3. Inferior subsegment of the lateral segment
  4. Superior and inferior subsegment of the medial segment
  5. Inferior subsegment of the anterior segment
  6. Inferior subsegment of the posterior segment
  7. Superior subsegment of the posterior segment
  8. Superior subsegment of the anterior segment
  %
    Whole liver | 13.7 (7.3) | 14.3 (7.9) | 14.0 (7.5)
    Couinaud Segment 1 | 13.1 (7.2) | 13.1 (7.3) | 13.1 (7.1)
    Couinaud Segment 2 | 12.9 (6.8) | 13.4 (7.7) | 13.1 (7.1)
    Couinaud Segment 3 | 13.5 (7.3) | 13.9 (7.7) | 13.7 (7.4)
    Couinaud Segment 4 | 13.4 (7.2) | 13.9 (7.6) | 13.6 (7.3)
    Couinaud Segment 5 | 13.9 (7.6) | 14.5 (8.3) | 14.1 (7.8)
    Couinaud Segment 6 | 13.6 (7.6) | 13.9 (8) | 13.7 (7.7)
    Couinaud Segment 7 | 13.9 (7.3) | 14.4 (7.8) | 14.1 (7.4)
    Couinaud Segment 8 | 14.0 (7.3) | 14.9 (8.1) | 14.4 (7.6)
Controlled attenuation parameter [Mean (Standard Deviation); unit: dB/m] — Controlled attenuation parameter (CAP) was measured by liver elastography, FibroScan.
  dB/m | 315.7 (43.9) | 320.2 (42.9) | 317.9 (43.1)
Liver stiffness [Mean (Standard Deviation); unit: kPa] — Liver stiffness was measured by liver elastography, FibroScan.
  kPa | 6.2 (1.8) | 5.8 (1.4) | 6.0 (1.7)
Comorbidities [Count of Participants; unit: Participants]
  Impaired glucose regulation | 16 | 20 | 36
  Type 2 diabetes | 14 | 10 | 24
  Hyperlipidaemia | 8 | 6 | 14
  Hypertension | 11 | 8 | 19
Concomitant drug use [Count of Participants; unit: Participants]
  Anti-lipidaemic | 4 | 2 | 6
  Anti-hypertensive | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change of Liver Fat Content in %
Description: Change of liver fat content in %.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: absolute fat content change in %
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
absolute fat content change in %
  Liver fat content measured by 1H-MRS | -20.5 [-25.0 to -15.9] | -15.5 [-20.3 to -10.8]
  Liver fat content measured by MRI-PDFF | -7.6 [-9.7 to -5.5] | -7.3 [-10.3 to -4.3]

2. Secondary Outcome: Change of Weight
Description: Change of weight in kilograms.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
kg | -5.3 [-6.4 to -4.2] | -3.8 [-5.0 to -2.6]

3. Secondary Outcome: Change of Blood Glucose: Fasting Blood Glucose
Description: Change of fasting blood glucose in mg/dL.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
mg/dL | -12.6 [-18.9 to -6.3] | -10.8 [-16 to -5.4]

4. Secondary Outcome: Change of Blood Glucose: 2h Postload Blood Glucose
Description: Change of 2h postload blood glucose in mg/dL.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
mg/dL | -50.6 [-67.9 to -33.3] | -71.6 [-94.9 to -48.6]

5. Secondary Outcome: Change of HbA1c
Description: Change of HbA1c in %.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: HbA1c in %
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
HbA1c in % | -0.5 [-0.7 to -0.3] | -0.1 [-0.2 to -0.02]

6. Secondary Outcome: Change of Liver Enzymes: Alanine Aminotransferase
Description: Change of alanine aminotransferase in U/L.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
U/L | -24.8 [-35.4 to -14.2] | -10.1 [-14.3 to -5.9]

7. Secondary Outcome: Change of Liver Enzymes: Aspartate Aminotransferase
Description: Change of aspartate aminotransferase in U/L.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
U/L | -11.5 [-17 to -5.9] | -4.3 [-6.8 to -1.8]

8. Secondary Outcome: Change of Liver Enzymes: γ-glutamyl Transpeptidase
Description: Change of γ-glutamyl transpeptidase in U/L.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
U/L | -16.5 [-25 to -8] | -6.3 [-12.3 to -0.3]

9. Secondary Outcome: Change of Lipid Profile: Total Cholesterol
Description: Change of total cholesterol in mg/dL.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
mg/dL | -3.9 [-13.9 to 6.2] | -4.6 [-13.1 to 3.9]

10. Secondary Outcome: Change of Lipid Profile: Triglyceride
Description: Change of triglyceride in mg/dL.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
mg/dL | -24.8 [-46 to -3.5] | -45.1 [-85.8 to -5.3]

11. Secondary Outcome: Change of Lipid Profile: High-density Lipoprotein-cholesterol
Description: Change of high-density lipoprotein-cholesterol in mg/dL.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
mg/dL | 5.8 [3.5 to 7.7] | 1.2 [-0.8 to 3.1]

12. Secondary Outcome: Change of Lipid Profile: Low-density Lipoprotein-cholesterol
Description: Change of low-density lipoprotein-cholesterol in mg/dL.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
mg/dL | -4.6 [-14.3 to 5] | 0.8 [-7.7 to 8.9]

13. Secondary Outcome: Change of Lipid Profile: Free Fatty Acid
Description: Change of free fatty acid in mg/dL.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
mg/dL | -1.7 [-4 to 0.3] | -1.4 [-3.1 to 0.3]

14. Other Pre Specified Outcome: Change of Fat Mass
Description: measured by bioimpedance analyzer, fat mass in kilograms.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
kg | -4.5 [-5.6 to -3.3] | -2.6 [-3.5 to -1.8]

15. Other Pre Specified Outcome: Change of Lean Mass
Description: measured by bioimpedance analyzer, skeletal muscle mass in kilograms.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
kg | -0.8 [-1.5 to -0.1] | -1 [-1.8 to -0.2]

16. Other Pre Specified Outcome: Change of Abdominal Adipose Tissue Area
Description: measured by MRI, including visceral adipose and subcutaneous adipose, all in square centimeter.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: square centimeter
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
square centimeter
  Visceral adipose area | -45.4 [-60.1 to -30.8] | -38.7 [-51.6 to -25.9]
  Subcutaneous adipose area | -43.9 [-63.2 to -24.6] | -30.4 [-52.3 to -8.4]

17. Other Pre Specified Outcome: Change of Liver Stiffness Measure of Liver Transient Elastography
Description: Change of liver stiffness measure of liver transient elastography, in kPa.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
kPa | -0.8 [-1.3 to -0.3] | -0.7 [-1.3 to -0.2]

18. Other Pre Specified Outcome: Change of Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) Index
Description: Change of HOMA-IR index from baseline to week 12. HOMA-IR index was calculated as fasting serum insulin (μU/ml) × fasting plasma glucose (mmol/l)/22.5. A HOMA-IR index higher than 75th quartile of non diabetes subjects is considered to be insulin resistance. However, due to differences in race, gender and research subjects, there is currently no recognized cut-off point. The cut-off values of HOMA-IR reported in previous studies varied greatly. A study on Caucasian non diabetes population showed that the cut-off value is 2.29. And a Chinese study proposed that the cut-off value of population over 40 years old in Shanghai was 4.31 for men and 4.51 for women.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: index
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
index | -2 [-3.2 to -0.8] | -1.6 [-2.7 to -0.4]

19. Other Pre Specified Outcome: Change of Fasting Insulin
Description: Change of fasting insulin in μU/mL.
Time Frame: From baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: μU/mL
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
Number analyzed (Participants) | 30 | 30
μU/mL | -5.3 [-8.7 to -1.8] | -3.7 [-7.5 to 0.2]

ADVERSE EVENTS:
Time Frame: From 1 to 12 weeks.
Description: No participant was at risk for Serious Adverse Events. No participant was at risk for All-Cause Mortality.
Arm/Group | Intermittent Calorie Restriction (ICR) | Control (Continuous Calorie Restriction, CCR)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 8/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent Calorie Restriction (ICR) (N=30) | Control (Continuous Calorie Restriction, CCR) (N=30)
Fatigue/Weakness (General disorders) | 5 (5) | 0 (0) — Fatigue/Weakness, mild, in fasting mimicking days of ICR group.
Dysphoria (General disorders) | 3 (3) | 0 (0) — Dysphoria, mild, in fasting mimicking days of ICR group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04283942/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT04283942/ICF_001.pdf